CLINICAL TRIAL: NCT02469532
Title: DANCE Partner: Inflammatory Biomarker Analysis by Femoropopliteal Revascularization Method and Treatment Outcomes
Status: Completed | Type: Observational
Sponsor: Mercator MedSystems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP0181
Record Dates: First submitted 2015-05-14; First posted 2015-06-11 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Angioplasty, Balloon

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Atherectomy: Up to 20 atherectomy procedures at up to 5 sites in the United States. Change in inflammatory biomarkers (hs-CRP, MCP-1 and MMP-9) from baseline to 24 hours post-procedure and 30-days post-revascularization procedure.
  This registry will also observe outcomes (target lesion revascularization rates, 6 and 12 month duplex ultrasound-detected binary restenosis with PSVR>2.4) post-atherectomy revascularization procedures.
  Interventions: Device: Atherectomy System
- Angioplasty: Up to 20 angioplasty procedures at up to 5 sites in the United States. Change in inflammatory biomarkers (hs-CRP, MCP-1 and MMP-9) from baseline to 24 hours post-procedure and 30-days post-revascularization procedure.
  This registry will also observe outcomes (target lesion revascularization rates, 6 and 12 month duplex ultrasound-detected binary restenosis with PSVR>2.4) post-angioplasty revascularization procedures.
  Interventions: Device: Balloon Angioplasty

INTERVENTIONS:
Device: Balloon Angioplasty — Device: Balloon Angioplasty Selection is driven by preference of the operator
  Groups: Angioplasty
Device: Atherectomy System — Device: Orbital or Directional or Laser Atherectomy Systems Atherectomy selection is driven by preference of the operator
  Groups: Atherectomy

SUMMARY:
This is a prospective, multi-center, observational registry to document the baseline, 24-hour and 30-day inflammatory response and procedural outcomes out to 12 month follow-up after femoropopliteal angioplasty or atherectomy-based revascularization procedures.

DETAILED DESCRIPTION:
This is a prospective, multi-center, observational registry to document the baseline, 24-hour and 30-day inflammatory response and procedural outcomes out to 12 month follow-up after femoropopliteal angioplasty or atherectomy-based revascularization procedures.

1. To observe the femoropopliteal revascularization outcomes post-angioplasty and/or atherectomy and to observe potential correlation between patency outcomes and the levels of MCP-1, C-reactive protein and MMP-9 from baseline to 24 hours and 30 days post-procedure.
2. To provide a comparator dataset to the investigational DANCE trial, which has the same enrollment criteria as this observational trial but includes the investigational use of a local drug therapy to limit inflammation caused by mechanical revascularization.

ELIGIBILITY:
Inclusion Criteria:

Screening Criteria

* Male or non-pregnant female ≥18 years of age
* Rutherford Clinical Category 2-4
* Clinical diagnosis of PAD requiring revascularization, secondary to atherosclerosis affecting a lower limb.
* Patient is willing to provide informed consent and comply with the required follow up visits Procedural Criteria
* De novo or nonstented restenotic lesions >90 days from prior angioplasty and/or atherectomy, at least 3 cm from any previously placed stent or vascular surgery site
* >70% diameter stenosis up to 15 cm in total length (with no greater than 3 cm length of contiguous intervening normal artery) in the superficial femoral and/or popliteal artery (between the profunda and tibioperoneal trunk)
* Reference vessel diameter ≥3mm and ≤ 8mm
* Successful wire crossing of lesion
* A patent artery proximal to the index lesion free from significant stenosis (significant stenosis is defined as >50% in iliac or >30% stenosis in common femoral artery) as confirmed by angiography (treatment of target lesion after successful treatment of iliac or common femoral artery lesions is acceptable)

Exclusion Criteria:

Screening Criteria

* Pregnant, nursing or planning on becoming pregnant in < 2years
* Life expectancy of <2 years
* Known active malignancy
* History of solid organ transplantation
* Patient actively participating in another investigational device or drug study
* History of hemorrhagic stroke within 3 months
* Previous or planned surgical or interventional procedure within 30 days of index procedure
* Chronic renal insufficiency with eGFR <29
* Prior bypass surgery, drug-coated balloon or stenting of the target lesion
* Contra-indication or known hypersensitivity to contrast media or physician prescribed antiplatelet regimen as applicable
* Systemic fungal infection
* Anticipated use of IIb/IIIa inhibitor prior to index lesion treatment
* Acute or sub-acute thrombus, acute vessel occlusion or sudden symptom onset
* Acute limb ischemia
* Inability to ambulate (e.g. from prior ipsilateral or contralateral amputation)
* Patient is receiving steroids already, however locally acting inhaled steroids for asthma treatment do not exclude patients from the trial Procedural Criteria
* Lesions extending into the trifurcation or above the profunda
* Heavy eccentric or moderate circumferential calcification at index lesion
* Lesion length is >15 cm as measured from proximal normal vessel to distal normal vessel, or there is no normal proximal arterial segment in which duplex ultrasound velocity ratios can be measured
* Inadequate distal outflow defined as absence of at least one patent tibial artery (no lesion >50% stenosis) with flow into the foot
* Use of adjunctive therapies other than angioplasty, atherectomy (mechanical or laser) or bare metal stenting (i.e. scoring/cutting balloon, drug-eluting stent, drug-coated balloon, cryoplasty, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female at least 18 years of age presenting with a de novo or nonstented restenotic lesions >90 days from prior angioplasty and/or atherectomy of lesions causing >70% narrowing in the superficial femoral and/or popliteal arteries and totalling up to 15 cm in length (with no greater than 3 cm length of contiguous intervening normal artery), Rutherford Category 2-4, and with a reference vessel diameter of 3 to 8 mm.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2015-05; Primary Completion 2017-10 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change in inflammatory biomarkers | Baseline to 24-hours post-procedure and 30-days post-procedure
  Change in inflammatory biomarkers (hs-CRP, MCP-1 and MMP-9) from baseline to 24 hours post-procedure and 30-days post-revascularization procedure.

SECONDARY OUTCOMES:
Target Lesion Revascularization | 6 and 12 months post-procedure
  This registry will prospectively collect data from patients diagnosed with peripheral arterial disease to observe the restenosis rates in peripheral arteries compared with subjects enrolled in the DANCE trial (Mercator MedSystems TSP0149).
Comparing biomarker (hs-CRP, MCP-1 and MMP-9) results | Baseline to 24 hours post-procedure and 30-days post-revascularization procedure
  This registry will prospectively collect data from patients diagnosed with peripheral arterial disease to observe the correlation between the levels of MCP-1, C-reactive protein and MMP-9 after angioplasty or atherectomy procedures in peripheral arteries compared with subjects enrolled in the DANCE trial (Mercator MedSystems TSP0149). Objective measurement of biomarkers will be performed by a contract laboratory to avoid bias.

CONTACTS AND LOCATIONS:
Overall Officials: Jason A Yoho, MD, Principal Investigator — Mission Research, New Braunfels, TX
Locations (6):
- United States (6):
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Endovascular Technologies (Willis Knighton Medical Center), Bossier City, Louisiana
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Rex Hospital, Raleigh, North Carolina
  - Mission Research Institute, New Braunfels, Texas
  - Palestine Regional Medical Center, Palestine, Texas